CLINICAL TRIAL: NCT05381571
Title: Integrating Reminiscence Technology Into Exercise Programs in Subacute Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Bruyere Academic Medical Organization (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bruyere
Record Dates: First submitted 2022-04-28; First posted 2022-05-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Rehabilitation
Keywords: Motivating Reminiscence Technology; Feasibility; Exercise Adherence

STUDY DESIGN:
Intervention Model Description: All recruited participants will use the reminiscence based physical therapy technology, three times weekly for a total of 12 weeks (average admission duration). The expected study enrolment period is 6 months to allow for multiple sets of participants to be recruited from the same medical unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reminiscence-based physical therapy (Experimental): Participants will use the reminiscence-based technology (jDome BikeAround) for 10-minute sessions for three times per week during the 12 week study enrolment period.
  Interventions: Other: Motivating reminiscence physical therapy

INTERVENTIONS:
Other: Motivating reminiscence physical therapy — The jDome BikeAround system involves participants using a stationary bike while their selected location is displayed in front of them on a domed projector screen using Google Street View. Using pedals on the bike they can propel themselves down the street, steer and change direction as they wish.

SUMMARY:
This study evaluates the feasibility of a randomized controlled trial to evaluate the impact of motivating reminiscence-based therapy on exercise adherence, mood and physical health within a subacute rehabilitation population. The jDome BikeAround technology displays user-specified Google Earth images onto a domed screen as the user pedals on a stationary bike, which fosters the experience of bicycling through that given environment. Participants will use the technology for 12 weeks during their regularly scheduled therapy sessions.

DETAILED DESCRIPTION:
Adherence to physical activity in older adults and those in a low-intensity rehabilitation program is important with respect to achieving the demonstrated benefits in mobility, physical function and overall health maintenance. Physical activities that incorporate motivational strategies can improve long-term adherence to therapy programs. The jDome BikeAround technology is one example, as it involves reminiscence therapy coupled with stationary bicycling. Participant's are able to visit any familiar locations or places they have wished to visit, thus providing a positive and interactive experience as they engage in physical activity.

Participants will be enrolled for a total of 12 weeks. They will have three 10 minute weekly sessions with the jDome BikeAround during their regularly scheduled therapy sessions. Feasibility will be evaluated by participant recruitment, program completion, rate of adverse events and staff acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the LIR (Low-intensity rehabilitation) or CMP (complex medical program) unit/floor where the research study is being conducted. Of note, both units receive low intensity rehabilitation services at baseline.
* Participants capable of providing informed consent or have a SDM capable of providing consent on their behalf
* Sufficient visual abilities to observe images on the domed screen
* Able to comprehend and communicate in English or French
* Minimum height requirement of 5'2" or 157cm in order to successfully fit the BikeAround system's stationary bike.

Exclusion Criteria:

* Physical limitations (as determined by the SVH healthcare/physiotherapy team) that prevent use of the jDome BikeAround. This includes:
* 1) Inability to coordinate/move lower limbs effectively to complete pedaling task
* 2) The pedaling exercise causes discomfort/pain greater than expected with physical activity
* 3) Medical treatment prevents usage of the system (i.e. continuous ventilatory needs for patients admitted within the CMP unit)
* Cognitive impairment (as determined by the SVH healthcare/physiotherapy team) that prevent use of the jDome BikeAround, such as:
* 1) Inability to sustain attention to focus on pedaling task
* 2) Inability to follow one-step commands.
* Known behavioral abnormalities (e.g. overly aggressive behavior) that in the opinion of the clinical care team might impede any meaningful participation in the project
* Those who are in the opinion of, the attending physician or clinical team, too unwell to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment | Baseline
  Determine the feasibility of a future randomized controlled trial to evaluate the impact of the jDome BikeAround system on exercise adherence, mood and physical health within a subacute rehabilitation population. Feasibility will be determined by the ability to recruit 60 participants (based on the average number of patients admitted to the rehab units).
Number of participants retained | Week 12
  Determine the feasibility of a future randomized controlled trial to evaluate the impact of the jDome BikeAround system on exercise adherence, mood and physical health within a subacute rehabilitation population. Feasibility will be determined by the number of sessions participants attended, out of the total number of sessions offered.
Rate of adverse events | Week 12
  The number of adverse events experienced by participants related to the use of the jDome BikeAround will be monitored to evaluate the feasibility of a future randomized controlled trial using this technology.
Staff Acceptance | Week 12
  Staff Acceptance will be determined by measuring the number of sessions staff assign participants to use the jDome BikeAround, out of their total number of therapy sessions (I.e. total sessions assigned to use jDome BikeAround out of total therapy sessions which is 3 weekly sessions x 12 weeks).

SECONDARY OUTCOMES:
Endurance | Total distance (meters) will be measured after each participant session (10 minutes) using the jDome BikeAround. This will occur 3 times per week throughout study duration for 12 weeks
  Total distance (meters) travelled during each jDome BikeAround therapy bike session.
Mood changes | Weekly after a jDome BikeAround session (for 12 weeks)
  Participant mood changes will be measured following their jDome BikeAround session using The Face Scale developed by Lorish and Maisiak (1986)
Functional Independence Measure (FIM score) | Baseline, week 6, week 12
  Standardized measure of disability used in rehabilitation populations. Measure evaluating 18 functional tasks on a scale of 1 (total care) to 7 (independent). Maximum 126 (best) and minimum is 18 (worst).
Satisfaction using jDome BikeAround - Participants | Baseline, week 6, week 12
  This measure will be assessed using semi-structured interviews
Satisfaction using jDome BikeAround - Staff | Baseline, week 6, week 12
  This measure will be assessed using online surveys for rehabilitation staff. 5-point scale from "strongly disagree, disagree, neutral, agree, strongly agree"
Emotional Impact | Baseline, week 6, week 12
  This measure will be assessed using semi-structured interviews with participants. This will assessed depending on participant verbal responses, not using any particular scale.
Impact on overall therapy experience - Participants | Baseline, week 6, week 12
  This measure will be assessed using semi-structured interviews with participants
Impact on overall therapy experience - Staff | Baseline, week 6, week 12
  This measure will be assessed using online surveys for rehabilitation staff. 5-point scale from "strongly disagree, disagree, neutral, agree, strongly agree"
Ease of instruction - Participants | Baseline, week 6, week 12
  This measure will be assessed using semi-structured interviews with participants
Ease of instruction - Staff | Baseline, week 6, week 12
  This measure will be assessed using online surveys for rehabilitation staff. 3 questions graded on a 5-point scale from "strongly disagree, disagree, neutral, agree, strongly agree"

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Vincent Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hay Group, HCC. Sub-Acute Care Capacity Plan. 2016.
- [Background] Foley N, McClure JA, Meyer M, Salter K, Bureau Y, Teasell R. Inpatient rehabilitation following stroke: amount of therapy received and associations with functional recovery. Disabil Rehabil. 2012;34(25):2132-8. doi: 10.3109/09638288.2012.676145. Epub 2012 Apr 23. PMID 22524794
- [Background] Dijkers MP, Zanca JM. Factors complicating treatment sessions in spinal cord injury rehabilitation: nature, frequency, and consequences. Arch Phys Med Rehabil. 2013 Apr;94(4 Suppl):S115-24. doi: 10.1016/j.apmr.2012.11.047. Epub 2013 Mar 7. PMID 23465468
- [Background] Laddu DR, Lavie CJ, Phillips SA, Arena R. Physical activity for immunity protection: Inoculating populations with healthy living medicine in preparation for the next pandemic. Prog Cardiovasc Dis. 2021 Jan-Feb;64:102-104. doi: 10.1016/j.pcad.2020.04.006. Epub 2020 Apr 9. No abstract available. PMID 32278694
- [Background] Lin YC, Dai YT, Hwang SL. The effect of reminiscence on the elderly population: a systematic review. Public Health Nurs. 2003 Jul-Aug;20(4):297-306. doi: 10.1046/j.1525-1446.2003.20407.x. PMID 12823790
- [Background] de Souto Barreto P, Rolland Y, Vellas B, Maltais M. Association of Long-term Exercise Training With Risk of Falls, Fractures, Hospitalizations, and Mortality in Older Adults: A Systematic Review and Meta-analysis. JAMA Intern Med. 2019 Mar 1;179(3):394-405. doi: 10.1001/jamainternmed.2018.5406. PMID 30592475
- [Background] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Background] Vogel T, Brechat PH, Lepretre PM, Kaltenbach G, Berthel M, Lonsdorfer J. Health benefits of physical activity in older patients: a review. Int J Clin Pract. 2009 Feb;63(2):303-20. doi: 10.1111/j.1742-1241.2008.01957.x. PMID 19196369
- [Background] American College of Sports Medicine Position Stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 1998 Jun;30(6):992-1008. PMID 9624662
- [Background] Rivera-Torres S, Fahey TD, Rivera MA. Adherence to Exercise Programs in Older Adults: Informative Report. Gerontol Geriatr Med. 2019 Jan 22;5:2333721418823604. doi: 10.1177/2333721418823604. eCollection 2019 Jan-Dec. PMID 30733977
- [Background] Mora JC, Valencia WM. Exercise and Older Adults. Clin Geriatr Med. 2018 Feb;34(1):145-162. doi: 10.1016/j.cger.2017.08.007. Epub 2017 Oct 10. PMID 29129214
- [Background] Ruano-Ravina A, Pena-Gil C, Abu-Assi E, Raposeiras S, van 't Hof A, Meindersma E, Bossano Prescott EI, Gonzalez-Juanatey JR. Participation and adherence to cardiac rehabilitation programs. A systematic review. Int J Cardiol. 2016 Nov 15;223:436-443. doi: 10.1016/j.ijcard.2016.08.120. Epub 2016 Aug 13. PMID 27557484
- [Background] Bredland EL, Soderstrom S, Vik K. Challenges and motivators to physical activity faced by retired men when ageing: a qualitative study. BMC Public Health. 2018 May 15;18(1):627. doi: 10.1186/s12889-018-5517-3. PMID 29764398
- [Background] Schutzer KA, Graves BS. Barriers and motivations to exercise in older adults. Prev Med. 2004 Nov;39(5):1056-61. doi: 10.1016/j.ypmed.2004.04.003. PMID 15475041
- [Background] Bennett JA, Winters-Stone K. Motivating older adults to exercise: what works? Age Ageing. 2011 Mar;40(2):148-9. doi: 10.1093/ageing/afq182. Epub 2011 Jan 20. No abstract available. PMID 21252038
- [Background] D'Cunha NM, Isbel ST, Frost J, Fearon A, McKune AJ, Naumovski N, Kellett J. Effects of a virtual group cycling experience on people living with dementia: A mixed method pilot study. Dementia (London). 2021 Jul;20(5):1518-1535. doi: 10.1177/1471301220951328. Epub 2020 Aug 21. PMID 32820955
- [Background] Huang HC, Chen YT, Chen PY, Huey-Lan Hu S, Liu F, Kuo YL, Chiu HY. Reminiscence Therapy Improves Cognitive Functions and Reduces Depressive Symptoms in Elderly People With Dementia: A Meta-Analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2015 Dec;16(12):1087-94. doi: 10.1016/j.jamda.2015.07.010. Epub 2015 Sep 1. PMID 26341034
- [Background] Cheng C, Fan W, Liu C, Liu Y, Liu X. Reminiscence therapy-based care program relieves post-stroke cognitive impairment, anxiety, and depression in acute ischemic stroke patients: a randomized, controlled study. Ir J Med Sci. 2021 Feb;190(1):345-355. doi: 10.1007/s11845-020-02273-9. Epub 2020 Jun 23. PMID 32578029
- [Background] Batchelor-Aselage M, Amella E, Zapka J, Mueller M, Beck C. Research with dementia patients in the nursing home setting: a protocol for informed consent and assent. IRB. 2014 Mar-Apr;36(2):14-20. No abstract available. PMID 24783377
- [Background] Lorish CD, Maisiak R. The Face Scale: a brief, nonverbal method for assessing patient mood. Arthritis Rheum. 1986 Jul;29(7):906-9. doi: 10.1002/art.1780290714. PMID 3741503